CLINICAL TRIAL: NCT02130687
Title: Contribution of Substance P to Blood Pressure Regulation in the Setting of Dipeptidyl Peptidase IV (DPP4) and Angiotensin-Converting Enzyme (ACE) Inhibition
Brief Title: Effect of Chronic ACE and DPP4 Inhibition on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, MD, Hugh Jackson Morgan Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 121253
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Results first posted 2021-07-26 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Type 2 Diabetes Mellitus; Hypertension; Angiotensin Converting Enzyme Inhibitors; Dipeptidyl Peptidase IV Inhibitors; Sitagliptin; Aprepitant; Ramipril
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — microcrystalline cellulose; Sitagliptin Phosphate; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amlodipine (Active Comparator): Subjects in this arm will receive calcium channel blocker therapy with amlodipine 5mg daily for 3 days then 10mg daily for 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Interventions: Drug: Placebo; Drug: Sitagliptin; Drug: Aprepitant; Other: Mixed Meal Test (MMT)
- Ramipril (Experimental): Subjects will receive ACE-inhibitor therapy with ramipril 5mg daily for 3 days, followed by 10mg daily for the remaining 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Interventions: Drug: Placebo; Drug: Sitagliptin; Drug: Aprepitant; Other: Mixed Meal Test (MMT)
- Valsartan (Active Comparator): Subjects will receive ARB therapy with valsartan 160mg daily for 3 days, followed by 320mg daily for the remaining 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Interventions: Drug: Placebo; Drug: Sitagliptin; Drug: Aprepitant; Other: Mixed Meal Test (MMT)

INTERVENTIONS:
Drug: Placebo — Subjects will receive two capsules of placebo to preserve the blinding of the study.
  In a separate period, subjects will receive one capsule of placebo and one capsule of sitagliptin.
  Other Names: Microcrystalline cellulose
Drug: Sitagliptin — Subjects will receive sitagliptin 100mg daily for 7 days. In addition, subjects will receive either aprepitant or a capsule of placebo to preserve the blinding of the study.
  Other Names: Januvia
Drug: Aprepitant — Subjects will receive aprepitant (125 mg on the first day followed by 80mg/d) for 7 days along with sitagliptin.
  Other Names: Emend
Other: Mixed Meal Test (MMT) — The first 18 subjects per arm/ group will undergo a mixed meal test on the 7th day of each medication intervention. This will take place after the first half of the study day at the clinical research center, following a 30 minute rest. Subjects will ingest a shake (combination of fixed carbohydrates/ fat/ protein) and have blood pressure, heart rate, and venous blood sample measurements collected for 4 hours after the meal.

SUMMARY:
In this study the investigators will test the hypothesis that dipeptidyl peptidase IV (DPP4) inhibition attenuates the antihypertensive effect of angiotensin-converting enzyme (ACE) inhibition but not angiotensin receptor blockade or calcium channel blockade. The investigators further hypothesize that this effect is mediated by substance P.

DETAILED DESCRIPTION:
The use of dipeptidyl peptidase IV (DPP4) inhibitors for the treatment of type 2 diabetes (T2DM) is growing rapidly. The majority of patients with T2DM are also taking ACE inhibitors or angiotensin receptor blockers (ARBs) in order to reduce cardiovascular and renal morbidity and mortality. DPP4 and ACE inhibitors share the common vasoactive substrate substance P. Substance P acts as a vasodilator but also activates the sympathetic nervous system. Understanding the interactive effects of DPP4 and ACE inhibitors on blood pressure and neurohumoral activation has important implications for the millions of patients with T2DM who take these drugs concurrently.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 80 years old

For female subjects the following conditions must be met:

Postmenopausal status for at least 1 year, or Status-post surgical sterilization, or If of childbearing potential, utilization of barrier methods of birth control and willingness to undergo urine β-HCG testing prior to drug treatment and on every study day

T2DM, as defined by 1 or more of the following at the time of screening visit:

* Hgb A1C ≥6.5%, or
* Fasting plasma glucose ≥126mg/dL, or
* 2-hour plasma glucose ≥200 mg/dL following 75gr oral glucose load

Hypertension, as defined by:

* Seated SBP ≥130 mm Hg on three occasions documented in medical record, or
* Seated DBP ≥80 mm Hg on three occasions documented in medical record, or
* Treatment with antihypertensive medications for a minimum of 6 months

Exclusion Criteria:

* Type 1 diabetes
* Poorly controlled T2DM, defined as Hgb A1C>8.7%
* Use of anti-diabetic medications other than metformin for at least 12 months prior to initiation of the study
* Secondary hypertension
* Subjects who have participated in a weight-reduction program during the last 6 months and whose weight has increased or decreased more than 5 kg over the preceding 6 months
* Pregnancy
* Breast-feeding
* Treatment with drugs primarily metabolized through CYP3A4 (e.g. cisapride, pimozide)
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy and diastolic dysfunction acceptable), deep vein thrombosis, pulmonary embolism, second- or third-degree AV block, mitral valve stenosis, or hypertrophic cardiomyopathy
* Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >3 x upper limit of normal range)
* Impaired renal function (eGFR< 50mL/min/1.73m2 as determined by the MDRD equation)
* History or presence of immunological or hematological disorders.
* History of pancreatitis or know pancreatic lesion
* History of angioedema while taking an ACE inhibitor
* Hematocrit <35%
* Treatment with anticoagulants
* Diagnosis of asthma requiring use of inhaled β-2 agonist more than 1 time per week
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Treatment with systemic glucocorticoids within the last 6 months
* Treatment with lithium salts
* Treatment with any investigational drug in the 1 month preceding the study
* Mental conditions rendering the subject unable to understand the nature, scope, or possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-06; Primary Completion 2020-05 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mashayekhi M, Wilson JR, Jafarian-Kerman S, Nian H, Yu C, Shuey MM, Luther JM, Brown NJ. Association of a glucagon-like peptide-1 receptor gene variant with glucose response to a mixed meal. Diabetes Obes Metab. 2021 Jan;23(1):281-286. doi: 10.1111/dom.14216. Epub 2020 Oct 22. PMID 33001556

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled if they met inclusion and exclusion criteria. 174 were consented to enroll 106. In other words, 68 of 174 consented were excluded because they did not meet inclusion/exclusion criteria.
Groups:
- Amlodipine: Subjects in this arm will receive calcium channel blocker therapy with amlodipine 5mg daily for 3 days then 10mg daily for 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Placebo: Subjects will receive two capsules of placebo to preserve the blinding of the study.
  In a separate period, subjects will receive one capsule of placebo and one capsule of sitagliptin.
  Sitagliptin: Subjects will receive sitagliptin 100mg daily for 7 days. In addition, subjects will receive either aprepitant or a capsule of placebo to preserve the blinding of the study.
  Aprepitant: Subjects will receive aprepitant (125 mg on the first day followed by 80mg/d) for 7 days along with sitagliptin.
  Mixed Meal Test (MMT): The first 18 subjects per arm/ group will undergo a mixed meal test on the 7th day of each medication intervention. This will take place after the first half of the study day at the clinical research center, following a 30 minute rest. Subjects will ingest a shake (combination of fixed carbohydrates/ fat/ protein) and have blood pressure, heart rate, and venous blood sample measurements collected for 4 hours after the meal.
- Ramipril: Subjects will receive ACE-inhibitor therapy with ramipril 5mg daily for 3 days, followed by 10mg daily for the remaining 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Placebo: Subjects will receive two capsules of placebo to preserve the blinding of the study.
  In a separate period, subjects will receive one capsule of placebo and one capsule of sitagliptin.
  Sitagliptin: Subjects will receive sitagliptin 100mg daily for 7 days. In addition, subjects will receive either aprepitant or a capsule of placebo to preserve the blinding of the study.
  Aprepitant: Subjects will receive aprepitant (125 mg on the first day followed by 80mg/d) for 7 days along with sitagliptin.
  Mixed Meal Test (MMT): The first 18 subjects per arm/ group will undergo a mixed meal test on the 7th day of each medication intervention. This will take place after the first half of the study day at the clinical research center, following a 30 minute rest. Subjects will ingest a shake (combination of fixed carbohydrates/ fat/ protein) and have blood pressure, heart rate, and venous blood sample measurements collected for 4 hours after the meal.
- Valsartan: Subjects will receive ARB therapy with valsartan 160mg daily for 3 days, followed by 320mg daily for the remaining 15 weeks. After 4 weeks of treatment, subjects will receive three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  Placebo: Subjects will receive two capsules of placebo to preserve the blinding of the study.
  In a separate period, subjects will receive one capsule of placebo and one capsule of sitagliptin.
  Sitagliptin: Subjects will receive sitagliptin 100mg daily for 7 days. In addition, subjects will receive either aprepitant or a capsule of placebo to preserve the blinding of the study.
  Aprepitant: Subjects will receive aprepitant (125 mg on the first day followed by 80mg/d) for 7 days along with sitagliptin.
  Mixed Meal Test (MMT): The first 18 subjects per arm/ group will undergo a mixed meal test on the 7th day of each medication intervention. This will take place after the first half of the study day at the clinical research center, following a 30 minute rest. Subjects will ingest a shake (combination of fixed carbohydrates/ fat/ protein) and have blood pressure, heart rate, and venous blood sample measurements collected for 4 hours after the meal.
Period: Washout
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 36 | 35 | 35
Completed | 36 | 33 | 31
Not Completed | 0 | 2 | 4
Period: Drug 1 Only
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 36 | 33 | 31
Completed | 33 | 30 | 30
Not Completed | 3 | 3 | 1
Period: Crossover Period 1
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 33 | 30 | 30
Completed | 33 | 30 | 30
Not Completed | 0 | 0 | 0
Period: Drug 1 Only Between Periods 1 and 2
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 33 | 30 | 30
Completed | 33 | 26 | 29
Not Completed | 0 | 4 | 1
Period: Crossover Period 2
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 33 | 26 | 29
Completed | 33 | 26 | 29
Not Completed | 0 | 0 | 0
Period: Drug 1 Only Between Periods 2 and 3
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 33 | 26 | 29
Completed | 33 | 25 | 27
Not Completed | 0 | 1 | 2
Period: Crossover Period 3
Arm/Group | Amlodipine | Ramipril | Valsartan
Started | 33 | 25 | 27
Completed | 33 | 25 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all participants who were randomized whether or not they received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine | Ramipril | Valsartan | Total
Number analyzed (Participants) | 36 | 35 | 35 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.9) | 52.9 (9.9) | 57.9 (10.4) | 56.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 17 | 53
  Male | 18 | 17 | 18 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 6 | 9 | 26
  White | 24 | 27 | 25 | 76
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 35 | 106

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure
Description: The primary analyses will focus on mean arterial blood pressure, heart rate, and norepinephrine (NE) concentrations during ramipril versus ramipril+sitagliptin, and during ramipril+sitagliptin versus ramipril+sitagliptin+aprepitant. We will make similar comparisons within the valsartan- and placebo-treated groups. In addition, we will compare blood pressure and heart rate parameters among the ramipril-treated, valsartan-treated, and placebo-treated groups during comparable concurrent treatment.
Time Frame: 4.5 hours on the 7th day of each intervention (placebo, sitagliptin, or sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Amlodipine Plus Placebo/Placebo: Participants received amlodipine 10mg/d for 15 weeks. During this intervention period they also received two placebo capsules for 7 days.
- Amlodipine Plus Sitagliptin/Placebo: Participants received amlodipine 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and a placebo capsule for 7 days.
- Amlodipine Plus Sitagliptin/Aprepitant: Participants received amlodipine 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and aprepitant 125mg/d for one day followed by 80 mg/d for a total of 7 days.
- Ramipril Plus Placebo/Placebo: Participants in this group received ramipril 10mg/d for 15 weeks. During this intervention period they also received two placebo capsules for one week for 7 days.
- Ramipril Plus Sitagliptin/Placebo: Participants in this group received ramipril 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and a placebo capsule.
- Ramipril Plus Sitagliptin/Aprepitant: Participants in this group received ramipril 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and aprepitant 125mg/d for one day followed by 80 mg/d for a total of 7 days.
- Valsartan Plus Placebo/Placebo: Participants in this group received valsartan 320mg/d for 15 weeks. During this intervention period they also received two placebo capsules for 7 days.
- Valsartan Plus Sitagliptin/Placebo: Participants in this group received valsartan 320mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and a placebo capsule for 7 days.
- Valsartan Plus Sitagliptin/Aprepitant: Participants in this group received valsartan 320mg/d for 15 weeks. During this intervention period they also received sitagliptin 100mg/day and aprepitant 125mg/d for one day followed by 80 mg/d for a total of 7 days.
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 33 | 33 | 33 | 27 | 25 | 28 | 28 | 29 | 29
mmHg | 94.42 (7.53) | 93.41 (8.75) | 91.54 (7.80) | 90.21 (12.46) | 89.88 (9.67) | 86.95 (10.16) | 94.54 (9.96) | 93.71 (10.75) | 93.98 (10.75)

2. Primary Outcome: Heart Rate
Description: The primary analyses will focus on blood pressure, heart rate, and norepinephrine (NE) concentrations during ramipril versus ramipril+sitagliptin, and during ramipril+sitagliptin versus ramipril+sitagliptin+aprepitant. We will make similar comparisons within the valsartan- and placebo-treated groups. In addition, we will compare blood pressure and heart rate parameters among the ramipril-treated, valsartan-treated, and placebo-treated groups during comparable concurrent treatment.
Time Frame: 4.5 hours on the 7th day of each intervention (placebo, sitagliptin, or sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 33 | 33 | 33 | 27 | 25 | 28 | 28 | 29 | 29
beats per minute | 69.59 (9.75) | 70.43 (9.79) | 69.41 (9.84) | 66.58 (7.71) | 66.30 (8.16) | 66.15 (8.06) | 66.19 (9.19) | 65.86 (8.46) | 65.10 (8.52)

3. Primary Outcome: Norepinephrine (NE) Concentrations
Description: as for outcome 2
Time Frame: 4.5 hours on the 7th day of each intervention (placebo, sitagliptin, or sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 32 | 32 | 32 | 27 | 25 | 27 | 28 | 28 | 28
pg/mL | 741.65 (660.82) | 730.88 (613.69) | 610.65 (587.19) | 470.69 (474.88) | 627.55 (593.92) | 649.39 (624.67) | 874.22 (863.75) | 986.31 (1114.67) | 1013.54 (1073.91)

4. Secondary Outcome: Low Frequency Variability of Blood Pressure Activity
Description: Low frequency variability of systolic blood pressure will be measured using spectral analysis.
Time Frame: for 5 minutes on the 7th day of each intervention (placebo, sitagliptin, sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: mmHg2
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 19 | 20 | 20 | 13 | 14 | 13 | 16 | 16 | 16
mmHg2 | 5.14 (2.65) | 7.32 (7.72) | 7.07 (6.57) | 8.78 (8.10) | 7.27 (5.91) | 12.18 (11.16) | 8.51 (5.43) | 7.81 (3.65) | 8.58 (6.57)

5. Secondary Outcome: Glucose
Description: measure of effectiveness of DPP4 inhibitor
Time Frame: fasting at 3 hours on the 7th day of each intervention (placebo, sitagliptin, sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 32 | 33 | 32 | 27 | 25 | 27 | 28 | 29 | 29
mg/dL | 123.78 (34.28) | 112.51 (29.96) | 109.08 (21.35) | 118.04 (21.79) | 107.55 (18.41) | 107.66 (17.47) | 112.01 (21.6) | 103.69 (18.13) | 99.75 (15.59)

6. Secondary Outcome: Insulin
Description: Measure of insulin resistance.
Time Frame: fasting insulin measured at 3 hours on the 7th day of each intervention (placebo, sitagliptin, sitatliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: microU/mL
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 26 | 22 | 21 | 21 | 21 | 22 | 20 | 21 | 20
microU/mL | 20.7 (10.36) | 20.72 (11.95) | 20.22 (16.32) | 26.15 (13.82) | 22.59 (13.01) | 26.02 (18.48) | 21.39 (16.22) | 19.92 (14.46) | 16.83 (10.58)

7. Secondary Outcome: Dipeptidyl Peptidase IV (DPP4) Activity
Description: Measure of DPP4 inhibitor administration.
Time Frame: for 4.5 hours on the 7th day of each intervention (placebo, sitagliptin, sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: nmol/mL/min
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 33 | 33 | 31 | 25 | 23 | 26 | 26 | 27 | 27
nmol/mL/min | 20.27 (6.80) | 7.34 (2.98) | 6.96 (4.33) | 20.61 (6.24) | 8.78 (6.5) | 7.71 (3.4) | 19.4 (7.14) | 7.83 (4.07) | 6.70 (3.53)

8. Secondary Outcome: Angiotensin Converting Enzyme (ACE) Activity
Description: This is a measure of activity of the angiotensin-converting enzyme (ACE). The assay is a kinetic assay (Labcore) that measures the rate of cleavage of an added ACE substrate over time and the results are reported in Units, which represent the rate of increase in fluorescent metabolite over 30 minutes under standard conditions at 37C.
Time Frame: for 4.5 hours on the 7th day of each intervention (placebo, sitagliptin, sitagliptin+aprepitant)
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 33 | 33 | 32 | 26 | 24 | 25 | 28 | 28 | 28
Units | 37.00 (14.56) | 40.15 (14.87) | 35.78 (13.73) | 15.44 (9.20) | 14.69 (9.37) | 13.46 (5.38) | 37.21 (14.75) | 36.68 (13.08) | 36.89 (13.20)

9. Secondary Outcome: Mean Arterial Blood Pressure
Description: Average of measurements made every five minutes beginning just prior to (time 0) and for four hours after the ingestion of a mixed meal
Time Frame: Value provided is the AVERAGE of measurements made every five minutes prior to (time 0) and for four four hours after ingestion of a mixed meal.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 20 | 20 | 20 | 15 | 15 | 15 | 16 | 16 | 16
mmHg | 96.0 (10.0) | 93.6 (8.9) | 92.9 (8.7) | 94.2 (11.3) | 92.6 (10.7) | 91.0 (9.6) | 94.2 (11.6) | 96.1 (8.8) | 94.5 (8.6)

10. Secondary Outcome: Heart Rate
Description: The average of measurements made every five minutes prior to (time 0) and for four four hours after ingestion of a mixed meal
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 20 | 20 | 20 | 15 | 15 | 15 | 16 | 16 | 16
bpm | 71.8 (13.1) | 70.3 (11.6) | 71.7 (13.0) | 69.9 (10.7) | 73.3 (9.2) | 72.0 (10.4) | 70.3 (11.9) | 71.9 (11.3) | 71.9 (11.3)

11. Secondary Outcome: Neuropeptide Y
Description: Measurement of Neuropeptide Y (NPY) concentrations
Time Frame: Neuropeptide Y concentration prior to ingestion of the mixed meal.
Measure: Mean (Standard Error); unit: pM
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 20 | 20 | 20 | 15 | 15 | 15 | 16 | 16 | 16
pM | 0.35 (0.28) | 0.52 (0.34) | 0.51 (0.33) | 0.32 (0.32) | 0.54 (0.26) | 0.52 (0.29) | 0.27 (0.15) | 0.50 (0.26) | 0.47 (0.28)

12. Secondary Outcome: 24hr Urinary Testing for Sodium
Description: Subjects will collect 24hr urine sample and bring with to the study day for analysis
Time Frame: Urine was collected for sodium for 24 hrs prior to each of the study days listed below. Study days occurred after each 7-day treatment arm (placebo/placebo, sitagliptin/placebo, or sitagliptin/aprepitant) within 3 anti-hypertensive groups.
Measure: Mean (Standard Deviation); unit: mEq
Arm/Group | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
Number analyzed (Participants) | 29 | 29 | 29 | 20 | 20 | 22 | 26 | 26 | 25
mEq | 147.66 (69.46) | 146.90 (74.29) | 154.42 (61.01) | 177.70 (74.48) | 162.05 (68.55) | 142.95 (94.62) | 158.77 (60.19) | 138.65 (44.48) | 160.92 (80.86)

13. Other Pre Specified Outcome: Aldosterone, Angiotensin II, and Plasma Renin Activity (PRA)
Description: renin-angiotensin system measurements were not done because there were not significant differences in blood pressure
Time Frame: for 4.5 hours on the 7th day of each intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion or for approximately 15 weeks.
Description: Information for adverse events are provided for each anti-hypertensive group. Most events occurred during periods before or between crossover treatment periods and these are listed as such.
Groups:
- Washout Prior to Amlodipine: Subjects in this arm received calcium channel blocker therapy with amlodipine 5mg daily for 3 days then 10mg daily for 15 weeks. Subjects underwent washout prior to starting amlodipine.
- Amlodipine Alone: Subjects in this arm received calcium channel blocker therapy with amlodipine 5mg daily for 3 days then 10mg daily for 15 weeks. After 4 weeks of treatment, subjects received three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions were: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  During the first four weeks and between crossover therapies, participants received amlodipine alone.
- Amlodipine Plus Sitagliptin/Placebo: Participants received amlodipine 10mg/d for 15 weeks. During this intervention period they also received two placebo capsules for 7 days.
- Amlodipine Plus Placebo/Placebo: Participants received amlodipine 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100 mg/day and a placebo capsule for 7 days.
- Amlodipine Plus Sitagliptin/Aprepitant: Participants received amlodipine 10mg/day for 15 weeks. During this intervention period they also received sitagliptin 100 mg/day and aprepitant 125 mg/d for one day followed by 80 mg/d for a total of 7 days.
- Washout Prior to Ramipril: Subjects received ACE-inhibitor therapy with ramipril 5mg daily for 3 days, followed by 10mg daily for the remaining 15 weeks. Subjects underwent washout prior to starting ramipril.
- Ramipril Alone: Subjects received ACE-inhibitor therapy with ramipril 5mg daily for 3 days, followed by 10mg daily for the remaining 15 weeks.
  After 4 weeks of treatment, subjects received three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions were: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  During the first four weeks and between crossover therapies, participants received ramipril alone.
- Ramipril Plus Placebo/Placebo: Participants in this group received ramipril 10mg/d for 15 weeks. During this intervention period they also received two placebo capsules for 7 days.
- Ramipril Plus Sitagliptin/Placebo: Participants in this group received ramipril 10mg/d for 15 weeks. During this intervention period they also received sitagliptin 100 mg/day and a placebo capsule for 7 days.
- Ramipril Plus Sitagliptin/Aprepitant: Participants in this group received ramipril 10mg/d for 15 days. During this intervention period they also received sitagliptin 100 mg/day and aprepitant 125 mg/d for one day followed by 80 mg/d for a total of 7 days.
- Washout Prior to Valsartan: Subjects received ARB therapy with valsartan 160mg daily for 3 days, followed by 320mg daily for the remaining 15 weeks. Subjects underwent washout prior to starting valsartan.
- Valsartan Alone: Subjects received ARB therapy with valsartan 160mg daily for 3 days, followed by 320mg daily for the remaining 15 weeks. After 4 weeks of treatment, subjects received three different 1 week concurrent interventions, in a cross-over fashion, separated by a 4 week washout. The interventions will be: placebo + placebo, sitagliptin + placebo, sitagliptin + aprepitant.
  During the first four weeks and between crossover therapies, participants received valsartan alone.
- Valsartan Plus Placebo/Placebo: Participants in this group received valsartan 320 mg/d for 15 weeks. During this intervention period they also received two placebo capsules for 7 days.
- Valsartan Plus Sitagliptin/Placebo: Participants in this group received valsartan 320 mg/d for 15 weeks. During this intervention period they also received sitagliptin 100 mg/day and a placebo capsule for 7 days.
- Valsartan Plus Sitagliptin/Aprepitant: Participants in this group received valsartan 320 mg/d for 15 weeks. During this intervention period they also received sitagliptin 100 mg/day and aprepitant 125 mg/d for one day followed by 80 mg/d for a total of 7 days.
Arm/Group | Washout Prior to Amlodipine | Amlodipine Alone | Amlodipine Plus Sitagliptin/Placebo | Amlodipine Plus Placebo/Placebo | Amlodipine Plus Sitagliptin/Aprepitant | Washout Prior to Ramipril | Ramipril Alone | Ramipril Plus Placebo/Placebo | Ramipril Plus Sitagliptin/Placebo | Ramipril Plus Sitagliptin/Aprepitant | Washout Prior to Valsartan | Valsartan Alone | Valsartan Plus Placebo/Placebo | Valsartan Plus Sitagliptin/Placebo | Valsartan Plus Sitagliptin/Aprepitant
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/33 | 0/33 | 0/33 | 0/35 | 0/33 | 0/27 | 0/25 | 0/28 | 0/35 | 0/31 | 0/28 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/33 | 0/33 | 0/33 | 0/35 | 0/33 | 0/27 | 0/25 | 0/28 | 1/35 | 1/31 | 0/28 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 4/36 | 1/36 | 7/33 | 4/33 | 9/33 | 3/35 | 3/33 | 3/27 | 1/25 | 4/28 | 5/35 | 0/31 | 4/28 | 5/29 | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Washout Prior to Amlodipine (N=36) | Amlodipine Alone (N=36) | Amlodipine Plus Sitagliptin/Placebo (N=33) | Amlodipine Plus Placebo/Placebo (N=33) | Amlodipine Plus Sitagliptin/Aprepitant (N=33) | Washout Prior to Ramipril (N=35) | Ramipril Alone (N=33) | Ramipril Plus Placebo/Placebo (N=27) | Ramipril Plus Sitagliptin/Placebo (N=25) | Ramipril Plus Sitagliptin/Aprepitant (N=28) | Washout Prior to Valsartan (N=35) | Valsartan Alone (N=31) | Valsartan Plus Placebo/Placebo (N=28) | Valsartan Plus Sitagliptin/Placebo (N=29) | Valsartan Plus Sitagliptin/Aprepitant (N=29)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
unstable angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — stenting
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Washout Prior to Amlodipine (N=36) | Amlodipine Alone (N=36) | Amlodipine Plus Sitagliptin/Placebo (N=33) | Amlodipine Plus Placebo/Placebo (N=33) | Amlodipine Plus Sitagliptin/Aprepitant (N=33) | Washout Prior to Ramipril (N=35) | Ramipril Alone (N=33) | Ramipril Plus Placebo/Placebo (N=27) | Ramipril Plus Sitagliptin/Placebo (N=25) | Ramipril Plus Sitagliptin/Aprepitant (N=28) | Washout Prior to Valsartan (N=35) | Valsartan Alone (N=31) | Valsartan Plus Placebo/Placebo (N=28) | Valsartan Plus Sitagliptin/Placebo (N=29) | Valsartan Plus Sitagliptin/Aprepitant (N=29)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/35 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2/31 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0/35 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0/31 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
edema (Vascular disorders) | 0 (0) | 0/35 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0/31 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0/35 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0/31 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
elevated blood pressure (Cardiac disorders) | 4 (4) | 0/35 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0/31 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
orthostasis (Cardiac disorders) | 0 (0) | 0/35 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1/31 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
hypokalemia (Renal and urinary disorders) | 0 (0) | 0/35 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0/31 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT02130687/Prot_SAP_ICF_000.pdf